CLINICAL TRIAL: NCT01480414
Title: Evaluation the Side Effects of Repeated Bone Marrow Derived Mono Nuclear Stem Cells Transplantation in Patients With Lower Limb Ischemic Ulcer
Brief Title: Side Effects of 4 Times Bone Marrow Mono Nuclear Transplantation in Patients With Ischemic Lower Limb
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Royan-PVD-002
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2010-07

CONDITIONS: Ischemic Ulcer
Keywords: bone marrow mono nuclear stem cell ischemic ulcer
MeSH Terms: interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 4times injection (Experimental): the patients with ischemic lower limb ulcer who underwent 4times stem cell injection.
  Interventions: Biological: 4times injection
- one injection (Experimental): Patients with peripheral artery disease underwent cell transplantation just one time.
  Interventions: Biological: stem cell transplantation

INTERVENTIONS:
Biological: 4times injection — bone marrow derived mono nuclear stem cell
  Arms: 4times injection
Biological: stem cell transplantation — Mono nuclear stem cell transplantation by intra muscular injection to the ischemic lower limb
  Arms: one injection

SUMMARY:
Critical limb ischemia (CLI) results from severe occlusive disease that impairs distal limb perfusion to the point where oxygen delivery is no longer adequate to meet the metabolic needs of the tissue, even under resting conditions. The limits of peripheral artery disease (PAD) compensatory mechanisms, such as distal vasodilatation and collateral formation, have been exceeded at this point. PAD is a widespread disease, affecting up to 15% of all adults older than 55 years. Formation of true new blood vessels, or angiogenesis, and development of collateral vessels from preexisting blood vessels, or arteriogenesis, is important in the pathophysiology of vascular disease. By stimulating these processes the investigators might be able to provide an alternative treatment strategy for patients with lower limb ischemia. In response to tissue injury and remodeling, neovascularization usually occurs via the proliferation and migration of progenitor endothelial cells (EPC) from preexisting vasculature. Indeed, recent studies have shown that bone-marrow mononuclear cell (BM-MNC) implantation increases collateral vessel formation in patients with limb ischemia. So the investigators determine to evaluate the efficacy of repeated MNC transplantation in patients with ischemic lower limb.

DETAILED DESCRIPTION:
In this study we transparent bone marrow derived mononuclear stem cells 4 times to the ischemic limb of 11 patients with PAD.first of all all the patients evaluate by physical examination,PFWD,ABI and serologic tests.then underwent bone marrow aspiration to take sample.In our lab the MNC are separated and divided in to equal doses.one of them inject to the ischemic foot and the othr one are freezed and inject after 3weeks.3 weeks after second injection again patient underwent bone marrow aspiration and the same process repeat.then after 4times transplantation,patients are followed up after 1,3,6,9,12 months after injection and evaluate by physical examination,PFWD,ABI and serologic tests.all the data are collected and analysed and the result will be shown.3 patients underwent cell transplantation just one time due to one time bone marrow aspiration.They are followed up after 1,3,6,9,12 months after injection and evaluate by physical examination,PFWD,ABI and serologic tests.at the end of the study patients with 4imes injection and 1time injection will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic lower limb based on TASK guide line
* Rutherford score:2,3
* ABI<0.6
* Absolute ankle pressure < 60 mmHg
* Both gender
* Age:20-62years

Exclusion Criteria:

* EF<30%
* Cr>2
* HbA1c>8%
* Bone marrow disorders:leukemia
* Cognitive disorders
* Infections
* MI with ST elevation during last month
* Malignancy
* Immunologic or rheumatologic disorders

Ages: 20 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
side effects | 3months
  evaluation the side effect of cell injection like:allergic reaction,fever,skin eruption,pain increasing,decrease in walking distance,ulcer severity

SECONDARY OUTCOMES:
PFWD | 3months
  Evaluation the pain free walking distance after cell transplantation.
ABI | 3months
  evaluation the improvement the score of ABI after stem cell transplantation .
size and depth of ulcer | 3months
  evaluation the improvement of ulcer by measuring the size and depth of ulcer in millimeter after transplantation.
Amputation | 6months
  Evaluation the need of limb amputation because of worsening the ulcer after cell injection.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; mohammad zafarghandi, MD, Study Director — surgery scientist; Nasser Aghdami, MD,PhD, Study Director — head of Royan cell therapy center; Behnam Molavi, MD, Principal Investigator — Surgery scientist
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- [Derived] Molavi B, Zafarghandi MR, Aminizadeh E, Hosseini SE, Mirzayi H, Arab L, Baharvand H, Aghdami N. Safety and Efficacy of Repeated Bone Marrow Mononuclear Cell Therapy in Patients with Critical Limb Ischemia in a Pilot Randomized Controlled Trial. Arch Iran Med. 2016 Jun;19(6):388-96. PMID 27293053